CLINICAL TRIAL: NCT00106626
Title: Phase I Clinical Trial of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With Pemetrexed and Cisplatin in Patients With Advanced Cancer
Brief Title: Suberoylanilide Hydroxamic Acid in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Executive Vice President, Clinical and Quantitative Sciences, Merck & Co., Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005_006; MK0683-012
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Results first posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-03

CONDITIONS: Advanced Cancer
Keywords: Advanced solid tumors including MPM and NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Pemetrexed; Cisplatin

ARMS (1):
- 1 (Experimental): vorinostat (Suberoylanilide Hydroxamic Acid [SAHA])
  Interventions: Drug: vorinostat (Suberoylanilide Hydroxamic Acid [SAHA]) in combination with Pemetrexed and Cisplatin

INTERVENTIONS:
Drug: vorinostat (Suberoylanilide Hydroxamic Acid [SAHA]) in combination with Pemetrexed and Cisplatin — Dose escalation study starting with vorinostat (Suberoylanilide Hydroxamic Acid [SAHA]) capsules 200 mg b.i.d. in combination with Pemetrexed and Cisplatin (see table for Reporting Groups).
  Other Names: MK0683; vorinostat; Suberoylanilide Hydroxamic Acid (SAHA)

SUMMARY:
The purpose of this investigational study is to determine the safety and tolerability of oral suberoylanilide hydroxamic acid when administered in combination with standard doses of pemetrexed and cisplatin for the treatment of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older with confirmed diagnosis of a solid tumor for which pemetrexed and cisplatin is acceptable treatment and have received no more than 2 prior systemic therapies
* Has at least 1 measurable lesion
* Has adequate blood, liver, and kidney functions
* Has not received any chemotherapy for at least 4 weeks prior to entry in this study
* Agrees to take adequate measures to prevent pregnancy as outlined in the protocol

Exclusion Criteria:

* Patient has been treated with other investigational agents with a similar anti-tumor mechanism
* Patient from Cohorts A and B has received pemetrexed or cisplatin within the past 6 months and from Cohorts C and D have received pemetrexed within the past 6 months
* Patient from Cohorts A and B has preexisting Grade 2 or higher neuropathy and from Cohorts C and D have Grade 3 or higher neuropathy
* Patient has active infection or had received IV (intravenous) antibiotic, antiviral, or antifungal medications within 2 weeks of the start of study drugs
* Patient has HIV, hepatitis B or hepatitis C infection
* Patient is pregnant or breast feeding
* Patient has allergy to any component of the study drugs
* Patient has history of GI (gastrointestinal) surgery or conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In = 29-Aug-05. Last Patient Last Visit = 03-Dec-07. Multicenter (4 Outpatient Clinics) in US.
Pre-assignment Details: Post-group assignment information: For all cohorts doses were administered in repeated 21-day cycles.
  Determination of the Maximum Tolerated Dose (MTD), by using dose-escalating design and measured by Dose Limiting Toxicity (DLT) is a standard procedure in the development of chemotherapeutic combinations.
Groups:
- Cohort A - Vorinostat BID + Pemetrexed + Cisplatin: Dose level A.1 - Vorinostat 200 mg twice daily (BID) for 14 days out of 3 weeks + Pemetrexed + Cisplatin
  Dose level A.2 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days in first week, two weeks off + Pemetrexed + Cisplatin
- Cohort B - Vorinostat QD + Pemetrexed + Cisplatin: Dose level B.1 - Vorinostat 300 mg once daily (QD) for 7 days + Pemetrexed + Cisplatin
  Dose level B.2 - Vorinostat 400 mg once daily (QD) for 7 days + Pemetrexed + Cisplatin
- Cohort C - Vorinostat BID + Pemetrexed: Dose level C.1 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days in first week, two weeks off + Pemetrexed
  Dose level C.2 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days in first two weeks, one week off + Pemetrexed
  Dose level C.3 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days repeated weekly + Pemetrexed
- Cohort D - Vorinostat QD + Pemetrexed: Dose level D.1 - Vorinostat 300 mg once daily (QD) for 7 days + Pemetrexed
  Dose level D.2 - Vorinostat 400 mg once daily (QD) for 7 days + Pemetrexed
Period: Overall Study
Arm/Group | Cohort A - Vorinostat BID + Pemetrexed + Cisplatin | Cohort B - Vorinostat QD + Pemetrexed + Cisplatin | Cohort C - Vorinostat BID + Pemetrexed | Cohort D - Vorinostat QD + Pemetrexed
Started | 13 | 9 | 14 | 16
Completed | 3 | 3 | 2 | 3
Not Completed | 10 | 6 | 12 | 13
Not completed — Adverse Event | 5 | 4 | 3 | 3
Not completed — Progressive Disease | 4 | 1 | 9 | 10
Not completed — Received radiation on new therapy | 1 | 0 | 0 | 0
Not completed — > 14 day delay in therapy start | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Vorinostat BID + Pemetrexed + Cisplatin | Cohort B - Vorinostat QD + Pemetrexed + Cisplatin | Cohort C - Vorinostat BID + Pemetrexed | Cohort D - Vorinostat QD + Pemetrexed | Total
Number analyzed (Participants) | 13 | 9 | 14 | 16 | 52
Age Continuous [Mean (Full Range); unit: years] | 60.52 [35 to 81] | 58.23 [31 to 74] | 60.09 [41 to 78] | 63.63 [39 to 81] | 61 [31 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 7 | 8 | 24
  Male | 9 | 4 | 7 | 8 | 28
Race/Ethnicity [Number; unit: participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black | 0 | 2 | 0 | 1 | 3
  European | 0 | 1 | 0 | 0 | 1
  Hispanic American | 1 | 0 | 0 | 2 | 3
  White | 12 | 6 | 14 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) Status as Determined by Number of Participants With Dose Limiting Toxicity (DLT) at Each Dose Level
Description: MTD was determined by the occurrence of DLTs during the first treatment cycle. DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. The dose level is equal to the MTD if < 2 patients experience a DLT and is also the highest tolerated dose level in the cohort.
Time Frame: Cycle 1 (21 days)
Population: A total of 52 participants were enrolled in this study. Six were violations pts (1 in Cohort C Dose Level 1, 1 in Cohort C Dose Level 2, 3 in Cohort D Dose Level 1, and 1 in Cohort D Dose Level 2) and were replaced. None of the violations pts had any DLTs in the first cycle of the study.
Measure: Number; unit: Participants
Groups:
- Dose Level A.1: (Cohort A) Dose level A.1 - Vorinostat 200 mg twice daily (BID) for 14 days out of 3 weeks + Pemetrexed + Cisplatin
- Dose Level A.2: (Cohort A) Dose level A.2 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days in first week, two weeks off + Pemetrexed + Cisplatin
- Dose Level B.1: (Cohort B) Dose level B.1 - Vorinostat 300 mg once daily (QD) for 7 days + Pemetrexed + Cisplatin
- Dose Level B.2: (Cohort B) Dose level B.2 - Vorinostat 400 mg once daily (QD) for 7 days + Pemetrexed + Cisplatin
- Dose Level C.1: (Cohort C) Dose level C.1 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days in first week, two weeks off + Pemetrexed
- Dose Level C.2: (Cohort C) Dose level C.2 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days in first two weeks, one week off + Pemetrexed
- Dose Level C.3: (Cohort C) Dose level C.3 - Vorinostat 300 mg twice daily (BID) for 3 consecutive days out of 7 days repeated weekly + Pemetrexed
- Dose Level D.1: (Cohort D) Dose level D.1 - Vorinostat 300 mg once daily (QD) for 7 days + Pemetrexed
- Dose Level D.2: (Cohort D) Dose level D.2 - Vorinostat 400 mg once daily (QD) for 7 days + Pemetrexed
Arm/Group | Dose Level A.1 | Dose Level A.2 | Dose Level B.1 | Dose Level B.2 | Dose Level C.1 | Dose Level C.2 | Dose Level C.3 | Dose Level D.1 | Dose Level D.2
Number analyzed (Participants) | 6 | 7 | 3 | 6 | 7 | 4 | 3 | 9 | 7
Participants
  Number (#) of DLT | 1 | 3 | 0 | 2 | 1 | 0 | 0 | 1 | 2
  # Participants treated at a dose level <MTD | 0 | 0 | 0 | 0 | 7 | 4 | 0 | 0 | 0
  # Participants treated at a dose level =MTD | 6 | 0 | 3 | 0 | 0 | 0 | 3 | 9 | 0
  # Participants treated at a dose level >MTD | 0 | 7 | 0 | 6 | 0 | 0 | 0 | 0 | 7

2. Secondary Outcome: Safety and Tolerability as Measured by the Number of Participants With Disease Progression
Description: Number of participants with disease progression (protocol-mandated reason for discontinuation). Disease progression was determined by the principle investigator.
Time Frame: Any time during 8 cycle treatment period through 30 days after.
Population: All participants. Treated Population includes all participants who received at least one dose and had efficacy measurements at baseline and at least one post baseline treatment.
Measure: Number; unit: Participants
Arm/Group | Cohort A - Vorinostat BID + Pemetrexed + Cisplatin | Cohort B - Vorinostat QD + Pemetrexed + Cisplatin | Cohort C - Vorinostat BID + Pemetrexed | Cohort D - Vorinostat QD + Pemetrexed
Number analyzed (Participants) | 13 | 9 | 14 | 16
Participants | 4 | 1 | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes